CLINICAL TRIAL: NCT06173388
Title: Efficacy of Structured Exercise Training Program on Swallowing and Ventilatory Functions in Patients With Cervicogenic Dysphagia
Brief Title: Exercise Training for Cervicogenic Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ashraf Abdelaal, Principal Investigator, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAPO-02-K-012-202
Record Dates: First submitted 2023-02-21; First posted 2023-12-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Dysphagia, Esophageal
Keywords: Deglutition Disorders; Pulmonary Functions; Manipulation; Physical Therapy
MeSH Terms: conditions — Deglutition Disorders | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The structured exercise training program (Experimental): Th study group received the structured exercise training program (composed of cervical stretching, strengthening and stabilizing exercises) plus the swallow resistance exercise.
  Interventions: Other: Structured exercise training program + The swallow resistance exercise program.; Other: Only the swallow resistance exercise program.
- The swallow resistance exercise (Other): The control group: received only the swallow resistance exercise.
  Interventions: Other: Only the swallow resistance exercise program.

INTERVENTIONS:
Other: Structured exercise training program + The swallow resistance exercise program. — Structured exercise training program + The swallow resistance exercise program.
  Other Names: Intervention for the study group.
  Arms: The structured exercise training program
Other: Only the swallow resistance exercise program. — Only the swallow resistance exercise program.
  Other Names: Intervention for the control group.

SUMMARY:
Background: Cervicogenic dysphagia is a swallowing difficulty caused by cervical problems that negatively impact pulmonary health, and quality of life and may increase the risk of mortality.

Study design: Randomized Controlled Study Purpose: The purpose was to explore the effect of a structured exercise training program composed of cervical stretching, strengthening and stabilizing exercises on the swallowing function, craniovertebral angle, and pulmonary function in patient with cervicogenic dysphagia.

Methods: 32 patients (age 35-50 years) with cervicogenic dysphagia were randomly allocated into study group (n=17) and control group (n=15). The craniovertebral angle (CVA), the swallowing function (using the swallow-difficulty questionnaire "SDQ") and the pulmonary function (including the forced vital capacity "FVC" and forced expiratory volume in one second "FEV1") were evaluated pre-study and post-study. All participants received three sessions/week for 8-weeks. The study group received the structured exercise program, in addition to the swallow resistance exercise (SRE), while the control group received the swallow resistance exercise only.

DETAILED DESCRIPTION:
Dysphagia is a common complaint in patients with cervical problems, and it is usually transient and responds favorably to rehabilitation programs. Cervicogenic dysphagia is difficulty in swallowing due to cervical spine pathology. Considering the close proximity of the cervical spine to the oropharynx and esophagus; the existence of any cervical pathology can adversely impact the pharynx and esophagus dimensions, through direct compression on the esophagus resulting in epiglottic tilt, cricopharyngeal spasm, and disturbed laryngeal inlet closure pattern, ending in disturbing the normal swallowing that can be evaluated by the swallowing disturbance questionnaire results in which the lower scores on the swallowing difficulty questionnaire reflects better swallowing status than higher scores, furthermore; with the cut-off value for 12.5 is a good predictor of the disturbed swallowing function.

Cervical malalignment is associated with an increased incidence of dysphagia. Cervical kyphosis is associated with malfunctional pharyngeal structure and disturbed swallowing. Additionally; cervical kyphosis is associated with deep cervical flexor muscles' weakness that in turn can significantly disturb cervical stability during swallowing. The combined effect of muscle weakness and poor cervical posture negatively impacts the laryngeal and cricopharyngeal sphincteric action and ends in cervical kyphosis.

Disturbed swallowing can negatively impact respiratory function, causing rapid deterioration in patients' ventilatory function and increasing the rate of pulmonary disorders' exacerbations. Maintaining normal swallowing function is essential in preventing consequent pulmonary complications.

Mal-aligned cervical spine predisposes to altered pulmonary functions that can be successfully corrected with therapeutic exercises, and manual therapy approaches.

A proper dysphagia management program is important not only to restore the normal coordinated swallowing-breathing pattern; but also, to eliminate the dysphagia-associated morbidity and health-related economic burden. Since cervicogenic dysphagia results from cervical spine pathologies or deformities, management of cervicogenic dysphagia should be focused on the treatment of cervical disturbances.

Postural correction therapeutic approaches are essential components in the dysphagia management program, but current evidence about their efficacy in dysphagia treatment is still limited. Although it is difficult to achieve a complete cervicogenic dysphagia cure; conservative therapies targeting postural realignment can alleviate the symptoms and treat cervicogenic dysphagia.

Definitely, there is a confirmed correlation between cervical spine pathologies and oropharyngeal dysphagia, further research is warranted to further explore the efficacy of the different rehabilitative non-surgical approaches in the treatment of cervicogenic dysphagia.

The objective of this study was to explore the efficacy of the structured physical therapy treatment program on pulmonary function, swallowing difficulty, and craniovertebral angle in patient with cervicogenic dysphagia.

ELIGIBILITY:
Inclusion Criteria:

Participants with cervicogenic dysphagia,

* Age 35-50 years,
* Patients with forward head posture (the craniovertebral angle ≤ 49 degree),
* Patients who agreed to sign the written consent.

Exclusion Criteria:

- Patients with unstable cardiopulmonary or psychological disorders.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Change from the baseline swallowing function at 8-weeks. | The swallowing function change was evaluated at the beginning of the study and after treatment completion (after 8 intervention weeks)
  The change in the swallowing function was evaluated across the 8 weeks period using the swallowing disturbance questionnaire. The swallowing function change was evaluated by assessing the swallowing function at the beginning of the study and at the end of the study (8 weeks interval).
  The swallowing disturbance questionnaire score greater than 12.5 indicates the presence of swallowing disturbances, with a high score reflecting increased dysphagia severity.
Change in the forward head position (through the craniovertebral angle value) was evaluated at 8-weeks. | The head position change was evaluated initially at the at beginning of the study and at the end of the study (8-weeks interval).
  The forward head position was evaluated across the 8-weeks period using the craniovertebral angle, defined between the horizontal line crossing the 7th cervical vertebra and second line extending from the 7th cervical vertebra to the ear tragus.
  The smaller craniovertebral angle is associated with greater forward head position, with the craniovertebral angle of ≤ 49 degrees suggesting the presence of forward head position.

SECONDARY OUTCOMES:
Change in the pulmonary functions | he pulmonary functions were evaluated initially at the at beginning of the study and at the end of the study (8-weeks interval).
  The pulmonary functions including the forced vital capacity and the forced expiratory volume in one second were evaluated using the portable spirometer.
  The pulmonary functions are usually expressed as percentages of predicted normal values %.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Abdelaal, Ph.D., Principal Investigator — Umm Al-Qura University
Locations (1):
- Umm Al-Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No